CLINICAL TRIAL: NCT00381407
Title: Organizational Skills Treatment for ADHD Children
Brief Title: Organizational Skills Training for Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Howard Abikoff, Director, Institute for Attention Deficit Hyperactivity and Behavior Disorders, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH074013 (NIH); R01MH074013 (NIH); DDTR B2-NDH
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Organizational Skills; Contingency Management
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will receive organizational skills training program
  Interventions: Behavioral: Organizational Skills Training
- 2 (Experimental): Participants will receive contingency management program
  Interventions: Behavioral: Contingency management (CM)
- 3 (No Intervention): Participants will receive wait list condition

INTERVENTIONS:
Behavioral: Organizational Skills Training — Participants in the OST group attend twenty 1-hour sessions over 10 weeks. OST trains children to use a variety of techniques for improving their organizational skills. Both children and their parents attend every OST session.
  Arms: 1
Behavioral: Contingency management (CM) — Participants in the CM group will attend twenty 1-hour sessions over 10 weeks. CM trains parents and teachers to identify desired "end" behaviors and to increase the frequency of these behaviors through the use of a structured reward system. Both children and their parents attend every CM session, but the children's participation will be minimal.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of organizational skills training in improving organizational, time management, and planning difficulties in children with attention deficit hyperactivity disorder.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common mental disorders among children. Children with ADHD frequently lack organizational, time management, and planning skills. These deficits can cause impaired functioning in multiple settings, including home, school, and peer relationships. Advancements in treatment options for these deficits, however, have been minimal. Previous research has indicated that organizational skills training (OST) is an effective intervention for improving organizational skills in children with ADHD. Its effectiveness relative to other available treatments is unknown. This study will compare the effectiveness of OST with that of contingency management (CM) and a waitlist condition in improving organizational, time management, and planning skills deficits in children with ADHD.

Participants in this study are randomly assigned to OST, CM, or Wait-List (WL). Participants in the OST and CM groups attend 20 1-hour sessions over 10 weeks. OST trains children to use a variety of techniques for improving their organizational skills. Both children and their parents attend every OST session. CM does not involve skills training. Rather, CM trains parents and teachers to identify desired "end" behaviors and to increase the frequency of these behaviors through the use of a structured reward system. Both children and their parents attend every CM session, but the children's participation will be minimal. Participants assigned to the waitlist condition will have the opportunity to receive their choice of either OST or CM once they have completed the study. All participants attend follow-up visits 1 month post-treatment. Participants assigned to OST and CM attend follow-up visits after 1 and 4 months into their next school grade. School performance, feelings about school, ADHD symptoms, organizational skills, family environment, medication or services received, and use of treatment strategies will be assessed at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Between grades 3 and 5 in school
* Meets criteria for ADHD, any subtype (a formal diagnosis prior to study entry is not necessary)
* Meets minimum score requirements on either Conners Parent or Conners Teacher Rating Scales
* Meets minimum criteria for organizational, time management, and planning deficits, as reported by parent or teacher
* Estimated IQ is greater than 85, as determined by the Wechsler Abbreviated Scale of Intelligence
* Has a teacher that is willing to participate
* Parents' schedule will allow attendance at study visits

Exclusion Criteria:

* Attends an all-day special education classroom or works with a para-professional in school
* Diagnosis of pervasive developmental disorder (PDD), psychosis, bipolar disorder, or post-traumatic stress disorder (PTSD)
* Current history of significant suicidality or sexual or physical abuse
* Any other comorbid psychiatric diagnosis or medical condition with significant symptoms that may interfere with study participation (e.g., severe depression, obsessive-compulsive disorder [OCD], or cystic fibrosis)
* Child's teacher has previously participated in this study

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Children's Organizational Skills Scale (COSS) | Measured immediatly post-treatment, Month 1 post-treatment, and Months 1 and 4 into the following school year
Academic Performance Rating Scale (APRS) | Measured immediatly post-treatment, Month 1 post-treatment, and Months 1 and 4 into the following school year

SECONDARY OUTCOMES:
Homework Problems Checklist | Measured immediatly post-treatment, Month 1 post-treatment, and Months 1 and 4 into the following school year
Family Environment Scale | Measured immediatly post-treatment, Month 1 post-treatment, and Months 1 and 4 into the following school year
Behavior Assessment System for Children | Measured immediatly post-treatment, Month 1 post-treatment, and Months 1 and 4 into the following school year

CONTACTS AND LOCATIONS:
Overall Officials: Howard B. Abikoff, PhD, Principal Investigator — New York University Child Study Center; Karen Wells, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - Duke University, Durham, North Carolina

REFERENCES:
- See also: Click here for the NYU Child Study Center website — http://www.aboutourkids.org